CLINICAL TRIAL: NCT05686252
Title: Investigating the Effect of Held Position During Kangaroo Care on Physiological Parameters of Premature Infants - A Randomised Controlled Trial
Brief Title: RCT: The Effect of Held Position During Kangaroo Care on Physiological Parameters of Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Cork University Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Professor, University College Cork
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 21121
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Extreme Prematurity; Extremely Low Birth Weight; Very Low Birth Weight Infant; Premature Birth
Keywords: Kangaroo Mother Care; NIRS; Oxygen saturation; Heart rate; NICU
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Superiority Crossover Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 degrees (Active Comparator): Baby is held at 30 degrees during kangaroo mother care in the NICU
  Interventions: Other: Held Position
- 60 degrees (Active Comparator): Baby is held at 60 degrees during kangaroo mother care in the NICU
  Interventions: Other: Held Position

INTERVENTIONS:
Other: Held Position — Change in angle of held position during kangaroo mother care to alternative angle

SUMMARY:
The goal of this superiority crossover randomised controlled trial is to investigate whether there is an optimal position at which to perform kangaroo mother care (KMC) in extremely preterm infants in the NICU. The main question it aims to answer is: 1) is there an optimal position for an infant to be held during KMC and 2) to optimise benefits for infants receiving KMC. Participants will be: 1) randomised into two groups which determine which angle they will start at first, 2) assessed over two hour-long sessions on different days with a change in the angle at the 30 minute point, 3) monitored using a Massimo NIRS machine which will record oxygen saturations, cerebral NIRS values and heart rates, and 4) monitored for any episodes of desaturations and bradycardias during this time. Participants will then be assessed beginning with the the other angle first on a different day. The researchers will then compare the two groups to see if being held at a 30 degrees during KMC is superior to being held at 60 degrees in terms of physiological stability.

DETAILED DESCRIPTION:
In this proposed study the investigators will examine whether there is an optimal position in which to perform KMC. This will be performed by evaluating cerebral oxygenation with near infrared spectroscopy (NIRS). Cerebral Near-Infrared Spectroscopy (NIRS) is used as a non-invasive assessment of cerebral oxygenation and cerebral hemodynamics. NIRS gives an estimation of the regional cerebral tissue oxygenation via a probe attached to the baby's forehead. It is minimally invasive and won't interrupt any of baby's cares or interrupt time with parents. The investigators will use NIRS to specifically examine whether there is a difference in physiological parameters between being held when the Mother/Father is at a 30 degree or 60 degree angle on the bedside recliner and whether better oxygenation is associated with one position over another. Currently there are no studies assessing the optimal position to carry out KMC in neonatal units. This study proposes to help answer a question which has not yet been answered in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Ex-premature infants who are a minimum of 28 weeks corrected gestational age
* Minimum weight at assessment for entry to study 600g
* Signed informed consent form

Exclusion Criteria:

* Corrected gestational age under 28 weeks
* Known neurological anomalies (not intraventricular Haemorrhage)
* Known orthopaedic conditions
* Known chromosomal anomalies

Min Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Mean cerebral NIRS values over KMC session | 2 hours in total per infant
  Mean cerebral NIRS values over the KMC session at the two different angles

SECONDARY OUTCOMES:
Mean peripheral saturation values over KMC session | 2 hours
  Mean peripheral saturation values over the KMC session at the two different angles
Mean heart rate values over KMC session | 2 hours
  Mean heart rate values over the KMC session at the two different angles
Number of bradycardias <100bpm over KMC session | 2 hours
  Number of bradycardias <100bpm over the KMC session at the two different angles
Number of Desaturations less than 80% for > 20 secs over KMC session | 2 hours
  Number of Desaturations less than 80% for > 20 secs over KMC session at the two different angles

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Maternity Hospital, Wilton, Cork, Munster, Ireland

REFERENCES:
- [Background] Ludington-Hoe SM, Johnson MW, Morgan K, Lewis T, Gutman J, Wilson PD, Scher MS. Neurophysiologic assessment of neonatal sleep organization: preliminary results of a randomized, controlled trial of skin contact with preterm infants. Pediatrics. 2006 May;117(5):e909-23. doi: 10.1542/peds.2004-1422. PMID 16651294
- [Background] Charpak N, Tessier R, Ruiz JG, Hernandez JT, Uriza F, Villegas J, Nadeau L, Mercier C, Maheu F, Marin J, Cortes D, Gallego JM, Maldonado D. Twenty-year Follow-up of Kangaroo Mother Care Versus Traditional Care. Pediatrics. 2017 Jan;139(1):e20162063. doi: 10.1542/peds.2016-2063. Epub 2016 Dec 12. PMID 27965377
- [Background] Jefferies AL; Canadian Paediatric Society, Fetus and Newborn Committee. Kangaroo care for the preterm infant and family. Paediatr Child Health. 2012 Mar;17(3):141-6. doi: 10.1093/pch/17.3.141. PMID 23449885
- [Derived] Stapleton I, Murphy S, Vaughan S, Walsh BH, Natchimuthu K, Livingstone V, Dempsey E. The effect of maternal position on cerebral oxygenation in premature infants during Kangaroo care: a randomised controlled trial. J Perinatol. 2025 Nov;45(11):1552-1557. doi: 10.1038/s41372-025-02287-0. Epub 2025 Apr 5. PMID 40186001